CLINICAL TRIAL: NCT04514523
Title: QBSAfe: A Novel Approach to Diabetes Management Focused on Quality of Life, Burden of Treatment, Social Integration and Avoidance of Future Events
Acronym: QBSAfe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Trinity Health Of New England (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000026483; 1R21AG061427-01 (NIH); 19-004560 (Other: Mayo)
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Results first posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Diabetes; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation Arm (Experimental)
  Interventions: Other: QBSAfe Toolkit

INTERVENTIONS:
Other: QBSAfe Toolkit — The QBSAfe toolkit focuses on palliating symptoms, alleviating burden of treatment, facilitating social connections, and optimizing treatment safety.

SUMMARY:
The purpose of this study is to co-develop a toolkit (known as the QBSAfe toolkit) with patients, family caregivers, and clinicians that focuses on palliating symptoms, alleviating burden of treatment, facilitating social connections, and optimizing treatment safety for patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

-Existing diagnosis of diabetes mellitus; have an existing appointment with a participating clinician

Exclusion Criteria:

* Do not speak English
* Severe vision/hearing impairment
* Unable to give informed consent for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Montori, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - Trinity Health of New England, Waterbury, Connecticut
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark JE, Boehmer KR, Breslin M, Haider S, Pasciak W, Gravholt D, Sanchez BB, Hartasanchez SA, El Kawkgi OM, Montori V, Lipska KJ. Quality of life, burden of treatment, safety, and avoidance of future events (QBSAfe) protocol: a pilot study testing an intervention to shift the paradigm of diabetes care. Pilot Feasibility Stud. 2021 Nov 8;7(1):196. doi: 10.1186/s40814-021-00935-8. PMID 34749816
- See also: Related Info — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-021-00935-8

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 84 participants and 7 clinicians
Groups:
- Single-Arm Intervention Group - Patients: QBSAfe Toolkit: The QBSAfe toolkit focuses on palliating symptoms, alleviating burden of treatment, facilitating social connections, and optimizing treatment safety.
- Single-Arm Intervention Group - Clinicians: Clinicians who participated in the study
Period: Overall Study
Arm/Group | Single-Arm Intervention Group - Patients | Single-Arm Intervention Group - Clinicians
Started | 84 | 7
Completed Video or Audio | 68 | 7
Completed Post Visit Questionnaire | 58 | 7
Completed | 58 | 7
Not Completed | 26 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were not collected for clinicians
Groups:
- Clinicians: Clinicians who participated in the study
- Total: Total of all reporting groups
Arm/Group | Implementation Arm | Clinicians | Total
Number analyzed (Participants) | 84 | 7 | 91
Age, Categorical [Count of Participants; unit: Participants] — Population: Baseline characteristics were not collected for clinicians
  Participants
    number analyzed (Participants) | 84 | 0 | 84
    <=18 years | 0 |  | 0
    Between 18 and 65 years | 39 |  | 39
    >=65 years | 45 |  | 45
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics were not collected for clinicians
  years
    number analyzed (Participants) | 84 | 0 | 84
    (all) | 74.4 (15.4) |  | 74.4 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics were not collected for clinicians
  Participants
    number analyzed (Participants) | 84 | 0 | 84
    Female | 39 |  | 39
    Male | 45 |  | 45
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics were not collected for clinicians
  Participants
    number analyzed (Participants) | 84 | 0 | 84
    American Indian or Alaska Native | 0 |  | 0
    Asian | 0 |  | 0
    Native Hawaiian or Other Pacific Islander | 0 |  | 0
    Black or African American | 14 |  | 14
    White | 66 |  | 66
    More than one race | 0 |  | 0
    Unknown or Not Reported | 4 |  | 4
Region of Enrollment [Number; unit: participants] — Population: Baseline characteristics were not collected for clinicians
  participants
    United States: number analyzed (Participants) | 84 | 0 | 84
    United States | 84 |  | 84

OUTCOME MEASURES:

1. Primary Outcome: Acceptability - Patients
Description: Patient responses to post-visit questionnaires.
Time Frame: Baseline [Post Clinical Encounter]
Population: Patients who had their visit recorded and answered post visit questionnaires
Measure: Count of Participants; unit: Participants
Groups:
- Single-Arm Intervention Group: QBSAfe Toolkit: The QBSAfe toolkit focuses on palliating symptoms, alleviating burden of treatment, facilitating social connections, and optimizing treatment safety.
Arm/Group | Single-Arm Intervention Group
Number analyzed (Participants) | 58
Participants
  These cards helped me talk about my situation during my visit: Strongly Agree | 16
  These cards helped me talk about my situation during my visit: Agree | 21
  These cards helped me talk about my situation during my visit: Neutral | 12
  These cards helped me talk about my situation during my visit: Disagree | 6
  These cards helped me talk about my situation during my visit: Strongly Disagree | 3
  I would like to have these cards available to me at my next visit: Strongly Agree | 12
  I would like to have these cards available to me at my next visit: Agree | 10
  I would like to have these cards available to me at my next visit: Neutral | 21
  I would like to have these cards available to me at my next visit: Disagree | 12
  I would like to have these cards available to me at my next visit: Strongly Disagree | 3
  I believe other patients like me would benefit from these cards: Strongly Agree | 19
  I believe other patients like me would benefit from these cards: Agree | 26
  I believe other patients like me would benefit from these cards: Neutral | 9
  I believe other patients like me would benefit from these cards: Disagree | 3
  I believe other patients like me would benefit from these cards: Strongly Disagree | 1

2. Primary Outcome: Acceptability - Clinicians
Description: Clinician responses to post-visit questionnaires.
Time Frame: Baseline [Post Clinical Encounter]
Population: Questionnaires completed by clinicians after each patient encounter
Measure: Count of Units; unit: Questionnaires after each encounter
Units Other Than Participants: Questionnaires after each encounter
Arm/Group | Single-Arm Intervention Group
Number analyzed (Participants) | 7
Number analyzed (Questionnaires after each encounter) | 69
Questionnaires after each encounter
  I felt confident in responding to issues raised by the patient: Strongly Agree | 48
  I felt confident in responding to issues raised by the patient: Agree | 14
  I felt confident in responding to issues raised by the patient: Neutral | 4
  I felt confident in responding to issues raised by the patient: Disagree | 3
  I felt confident in responding to issues raised by the patient: Strongly Disagree | 0
  I would like to use these cards with a patient like this next time: Strongly Agree | 43
  I would like to use these cards with a patient like this next time: Agree | 11
  I would like to use these cards with a patient like this next time: Neutral | 14
  I would like to use these cards with a patient like this next time: Disagree | 1
  I would like to use these cards with a patient like this next time: Strongly Disagree | 0
  I would recommend these cards to my colleagues: number analyzed (Questionnaires after each encounter) | 68
  I would recommend these cards to my colleagues: Strongly Agree | 46
  I would recommend these cards to my colleagues: Agree | 10
  I would recommend these cards to my colleagues: Neutral | 11
  I would recommend these cards to my colleagues: Disagree | 1
  I would recommend these cards to my colleagues: Strongly Disagree | 0

3. Secondary Outcome: Feasibility 1
Description: Percentage of participants who completed the study procedures.
Time Frame: Baseline [Post Clinical Encounter]
Population: Number of patients and number of clinicians in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm Intervention Group - Patients | Single-Arm Intervention Group - Clinicians
Number analyzed (Participants) | 84 | 7
Participants | 58 | 7

4. Secondary Outcome: Feasibility 2
Description: Percentage of recorded visits in which the QBSAFE toolkit was used assessed by Number of visits QBSAFE was used/Number of recorded visits.
Time Frame: Baseline [Post Clinical Encounter]
Measure: Number; unit: percentage of visits QBSAFE was used
Arm/Group | Implementation Arm
Number analyzed (Participants) | 58
percentage of visits QBSAFE was used | 58

5. Secondary Outcome: Feasibility 3
Description: Time to recruit 84 subjects across 3 sites.
Time Frame: Baseline [Post Clinical Encounter]
Population: Number of recruited patients
Measure: Number; unit: Days
Arm/Group | Implementation Arm
Number analyzed (Participants) | 84
Days | 145

ADVERSE EVENTS:
Time Frame: Up to 1 week.
Description: Study took place during routine clinical encounters. A subgroup of participants were followed for up to a week to complete qualitative interviews. Adverse events were not tracked for clinician arm.
Groups:
- Clinicians: Clinicians who participated in study
Arm/Group | Single-Arm Intervention Group | Clinicians
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/0
Other Adverse Events (participants affected / at risk) | 0/84 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT04514523/Prot_000.pdf